CLINICAL TRIAL: NCT03870945
Title: A Phase I/II Safety, Dose Finding and Feasibility Trial of MB-CART2019.1 in Patients With Relapsed or Resistant B-NHL
Brief Title: Safety of MB-CART2019.1 in Lymphoma Patients (MB-CART2019.1 Lymphoma / DALY 1)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2018-331
Record Dates: First submitted 2019-02-25; First posted 2019-03-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: B-cell Non Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose level 1 with 1x10^6 MBCART2019.1 per kg BW (Experimental): The IMP will be administered as an intravenous infusion. This is a 6+3 trial arm with 1x10^6 MBCART2019.1 per kg BW in a single infusion. If none or one of the six patients at dose level 1 experiences a dose limiting toxicity, another six patients will be treated at dose level 2. If two DLTs are observed at dose level 1 another three patients will be treated with the same dose. Dose escalation continues until at least >2 patients among a cohort of six to nine patients experience dose-limiting toxicities or dose level 2 is completed. The MTD is defined as the dose level below the dose inducing a DLT in more than 2 patients within one dose level.
  Interventions: Biological: MB-CART2019.1 Dose level 1
- Dose level 2 with 2.5x10^6 MBCART2019.1 per kg BW (Experimental): The IMP will be administered as an intravenous infusion. This is a 6+3 trial arm with 2.5x10^6 MBCART2019.1 per kg BW in a single infusion and maximum 2 dose levels. If none or one of the six patients at dose level 1 experiences a dose limiting toxicity, another six patients will be treated at dose level 2. If two DLTs are observed at dose level 1 another three patients will be treated with the same dose. If more than two DLTs are observed at dose level 1, trial will continue at dose level 0. Dose escalation continues until at least >2 patients among a cohort of six to nine patients experience dose-limiting toxicities or dose level 2 is completed. The MTD is defined as the dose level below the dose inducing a DLT in more than 2 patients within one dose level.
  Interventions: Biological: MB-CART2019.1 Dose level 2

INTERVENTIONS:
Biological: MB-CART2019.1 Dose level 1 — This is a prospective, multi-center, open phase I/II trial to evaluate feasibility, dosage, safety and toxicity as well as efficacy of ex vivo expanded autologous T cells genetically modified to express anti-CD20 and CD19 immunoreceptor (MBCART2019.1) in patients with relapsed or resistant aggressive CD20 and CD19 positive B-NHL/CLL/SLL.
  Other Names: CD2019-targeting CAR T cells; Anti-CD2019 CAR T cells
  Arms: Dose level 1 with 1x10^6 MBCART2019.1 per kg BW
Biological: MB-CART2019.1 Dose level 2 — This is a prospective, multi-center, open phase I/II trial to evaluate feasibility, dosage, safety and toxicity as well as efficacy of ex vivo expanded autologous T cells genetically modified to express anti-CD20 and CD19 immunoreceptor (MBCART2019.1) in patients with relapsed or resistant aggressive CD20 and CD19 positive B-NHL.
  Other Names: CD2019-targeting CAR T cells; Anti-CD2019 CAR T cells
  Arms: Dose level 2 with 2.5x10^6 MBCART2019.1 per kg BW

SUMMARY:
This is a prospective, multi-center, open phase I/II trial to evaluate feasibility, dosage, safety and toxicity as well as efficacy of ex vivo expanded autologous T cells genetically modified to express anti-CD20 and CD19 immunoreceptor (MBCART2019.1) in patients with relapsed or resistant aggressive CD20 and CD19 positive B-NHL/CLL/SLL.

DETAILED DESCRIPTION:
This trial will be performed as a multi-center phase I/II trial with MB-CART2019.1 and consists of part I. In part I, 12 to 18 patients with relapsed or resistant CD20 and CD19 positive NHL/CLL/SLL will be treated. Six plus three (6+3) patients in dose level 1 and 2 will be treated.

The trial will be conducted in Hematology Departments of Hospitals which meet the structural and personnel requirements for performing the planned regular trial-related investigations. Only sites will be chosen with expertise in and necessary facilities for managing cytokine release storm and other severe adverse events associated with this therapy such as neurotoxicity. A corresponding training to site personnel prior to trial start must be performed. The responsible intensive care unit (ICU) must be informed about the clinical trial before inclusion of the first patient and the respective dosing date in order to make sure that the medical staff of the ICU is able to react appropriately without any loss of time in case of emergency. The University Hospital of Cologne will provide the Coordinating Investigator. Additional clinical sites may be added during the trial.

Patients will be screened between day -30 and day -15. If the patient satisfies all the protocol inclusion and none of the exclusion criteria, he/she will be included in the clinical trial. Leukapheresis will be performed at the collection center on day -14 according to local standard practice. The leukapheresis product of the patient will be shipped by a special courier to the designated manufacturing center assigned by the sponsor. The leukapheresis sample will be used for the individual manufacturing of MB-CART2019.1 by using the automated CliniMACS Prodigy® System. The manufacturing of MB-CART2019.1 will start on day -13 and will be finished on day -1.

On day 5 of the manufacturing process the IPC (in-process-control) will indicate, if the manufacturing process is successful. Therefore, the lymphodepleting chemotherapy must only be started after the positive result of the IPC was confirmed by the manufacturer. Chemotherapy for lymphodepletion will be done on days -5 to -3.

Administration of MB-CART2019.1 will be performed on day 0 in the Hematology Departments of all sites. Patients will be followed up as inpatients until week 4 with close monitoring of their vital functions and lab parameters for signs of adverse events. In the second follow-up phase (week 4 until week 12), response will be assessed, and adverse events will be documented. A follow-up examination will be performed at week 12 (achievement of primary endpoint) and at month 12 which is considered end of trial or end of active part of the trial. In the long-term follow-up yearly until 5 years or patient's death, safety and response assessment as well as persistence of MBCART2019.1 will be performed. These assessments will be analyzed and reported separately and are not part of the entire clinical trial. This is a 6+3 trial design with a 0.3 log dose increment (1x106/2.5x106 MBCART2019.1 per kg BW in a single infusion) and maximum 2 dose levels. If none or one of the six patients at dose level 1 experiences a dose limiting toxicity, another six patients will be treated at dose level 2. If two DLTs are observed at dose level 1 another three patients will be treated with the same dose. If more than two DLTs are observed at dose level 1, trial will continue at dose level 0. Dose escalation continues until at least >2 patients among a cohort of six to nine patients experience dose-limiting toxicities or dose level 2 is completed. The MTD is defined as the dose level below the dose inducing a DLT in more than 2 patients within one dose level. DLT will be evaluated within 4 weeks after the infusion of MB-CART2019.1. An interval of at least 28 days between the treatment of the first and the second patient in each dose level is mandatory. An observation period for DLT of 28 days is considered to be safe to exclude potential toxicities prior to inclusion of the next patients into the same dose group or prior to dose escalation.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory/relapsed B-NHL (including malignant transformation like Richter's transformation) with no available approved standard therapy. Including, but not restricted to:

   1. Diffuse large B cell lymphoma (DLBCL): relapsed/refractory disease after ASCT or ineligible for ASCT after first-line therapy; transformation from CLL, SLL or FL allowed
   2. Follicular lymphoma: at least 2 prior regimens and progression <2 years after most recent line of therapy
   3. Mantle cell lymphoma: beyond 1st CR with relapsed disease, progressive disease during first-line rituximab chemotherapy, or persistent disease after first-line rituximab-chemotherapy and not eligible or appropriate for conventional therapy, ASCT or relapsed after prior autologous SCT, prior therapies including ibrutinib if not contraindicated
   4. CLL and SLL: after at least two lines of treatment including btk inhibitor ibrutinib and bcl2 inhibitor venetoclax (if not contraindicated), patients must have been refractory to at least one of the substances

   Patients with criteria 1b-d will only be eligible for Part I, dose cohort 1.
2. Patients in cohort 1a must have histologically confirmed DLBCL and associated subtypes with relapse or refractory disease after first line chemo-immunotherapy and be ineligible for HSCT
3. Histologically confirmed DLBCL and associated subtypes, defined by WHO 2016 classification:

   * DLBCL not otherwise specified (NOS)
   * High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements with DLBCL histology (DHL/THL) and FL3B
   * Aggressive B-cell lymphoma
   * T-cell/histocyte rich B-cell lymphoma
   * Primary mediastinal B-cell lymphoma
   * EBV+ DLBCL
   * Transformed lymphoma (e.g. transformed follicular or marginal zone lymphoma)
4. First line chemo-immunotherapy is defined as therapy containing the combination of CD20 targeted immunotherapy and cytotoxic chemotherapy.
5. Chemotherapy-refractory disease is defined as one or more of the following:

   * No response to first line of therapy

     * PD as best response to first line therapy regimen
     * SD as best response after 4 cycles of first line therapy
   * Disease progression or relapsed ≤12 months of first line therapy (must have biopsy proven recurrence in relapsed individuals)
6. Ineligibility for HSCT is defined as having ONE of the following criteria:

   * Age based on country-specific definition
   * Impaired pulmonary function (DLCO or FEV1 ≤60%)
   * Impaired cardiac function (LVEF <50%)
   * Impaired renal function (CrCl <60 mL/min)
   * Impaired hepatic function (AST/ALT >3 x ULN, bilirubin >1.5 x ULN or patient's baseline)

   In addition, all patients must fulfil the following criteria:
7. Age ≥18 years
8. Measurable disease according to Lugano criteria
9. CD19 or CD20 tumor expression is not required after first line chemo-immunotherapy.

   1. Must have archival tissue available, if received CD19 targeted therapy or CD20 antibody, archival tissue must have been obtained subsequent to that therapy
   2. Must have at least 10 unstained slides of tissue available
   3. If archival tissue is not available, must be willing to undergo attempted repeat biopsy and fine needle Aspiration
10. If has history of CNS disease, then must have:

    1. No signs or symptoms of CNS disease
    2. No active disease on magnetic resonance imaging (MRI)
    3. Absence of large cell lymphoma in cerebral spinal fluid (CSF) on cytospin preparation and flow cytometry, regardless of the number of white blood cells
11. If has history of cerebral vascular accident (CVA):

    1. The CVA event must be >12 months prior to leukapheresis
    2. Any neurological deficits must be stable
12. Estimated life expectancy of >3 months other than primary disease
13. No childbearing potential (i.e. postmenopausal, absence of menstrual bleeding for at least 1 year), hysterectomy, bilateral ovariectomy or tubal section/ligation) or negative pregnancy test at screening and before chemotherapy in women of childbearing potential. Sexually active female patients of childbearing potential should use one of the following highly effective methods of contraception (Pearl index <1%): hormonal contraceptives (oral, injected, implanted, transdermal), intrauterine devices or systems (e.g. hormonal and non-hormonal IUD), or vasectomized sexual partner for at least 1 month before the trial start, during the trial and in the 6 months following dosing. Male patients, unless surgically sterile (meaning at least two consecutive analyses following vasectomy demonstrate absence of sperms in the ejaculate), must be using two acceptable methods for contraception (e.g. spermicide and condom) during the trial and refrain from fathering a child throughout the trial and for up to 12 months after dosing
14. Signed and dated informed consent before conduct of any trial-specific procedure

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) performance status >2
2. Absolute neutrophil count (ANC) <1,000/µL
3. Platelet count <50,000/µL
4. Absolute lymphocyte count <100/µL
5. Presence of leukemia/lymphoma cells in peripheral blood
6. Primary CNS lymphoma
7. Unable to give informed consent
8. Known history of infection with human immunodeficiency virus (HIV) or active infection with hepatitis B (HGsAg positive)
9. Known history of infection with hepatitis C virus unless treated and confirmed to be polymerase chain reaction (PCR) negative
10. Known history or presence of seizure activities or on active anti-seizure medications within the previous 12 months
11. Known history of CVA within prior 12 months
12. Known history or presence of autoimmune CNS disease, such as multiple sclerosis, optic neuritis or other immunologic or inflammatory disease
13. Presence of CNS disease that, in the judgment of the investigator, may impair the ability to evaluate neurotoxicity
14. Active systemic fungal, viral or bacterial infection
15. Clinical heart failure with New York Heart Association class ≥2 or LVEF <30%
16. Resting oxygen saturation <90% on room air
17. Liver dysfunction as indicated by total bilirubin, AST and/or ALT >5 x institutional ULN, unless directly attributable to patient's tumor
18. CrCl <30 mL/min calculated according to the modified formula of Cockcroft and Gault or by direct urine collection
19. Pregnant or breast-feeding woman
20. Active secondary malignancy requiring treatment
21. Medical condition requiring prolonged use of systemic corticosteroids >10 mg/day
22. Concurrent radiotherapy (allow up to time of leukapheresis)
23. Baseline dementia that would interfere with therapy or monitoring, determined using mini-mental status exam at baseline
24. History of severe immediate hypersensitivity reaction against any drug or its ingredients/impurities that is scheduled to be given during trial participation e.g. as part of the mandatory lymphodepletion protocol, premedication for infusion, or rescue medication/salvage therapies for treatment related toxicities
25. Patients in which such medication (see exclusion criterion 24) is contraindicated for other reasons than hypersensitivity (e.g. live vaccines and fludarabine)
26. Refusal to participate in CAR-T long-term follow-up (LTFU).
27. Refusal to undergo core needle biopsy or fine needle aspiration of tumor on day 2-5 after MB-CART infusion and at time of disease progression and relapse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2024-05-28 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose of MB-CART2019.1 | Day 28 after infusion of MB-CART2019.1
  Determination of the MTD, defined as the highest dose level at which <33% of patients experience DLT until day 28 after infusion of MB-CART2019.1 or 2.5x106 MB-CART2019.1 per kg BW, whichever occurs first.
Safety and toxicity assessment of MB-CART2019.1 | Day 28 after infusion of MB-CART2019.1
  Safety and toxicity assessment per AE reporting classified according to CTCAE Version 5.

SECONDARY OUTCOMES:
Preliminary evidence of response to treatment | Weeks 4, 12, months 6 and 12 after infusion of MB-CART2019.1
  Objective response rate: (sum of CR+PR), CR, PR, SD and PD is defined according to Lugano criteria (DLBCL, FL. MCL) or IWCLL criteria (CLL/SLL)
Phenotype and persistence of MB-CART2019.1 | Days 2, 6, 9; Weeks 2, 3, 4, 6, 8, 12, months 6, 9, and 12 after infusion of MB-CART2019.1
  Blood samples for determination of persistence/phenotyping of infused MB-CART2019.1 will be analysed
Overall Survival | 12 months after infusion of MB-CART2019.1
  Determination of Overall Survival rate (OS) after Infusion of MB-CART2019.1
Best Overall Response (BOR) | Weeks 4 + 12, months 6 + 12 after infusion of MB-CART2019.1
  Best Overall Response recorded to study treatment after infusion of MB-CART2019.1 per Investigator assessment
Occurence of B-cell aplasia | weeks 2, 4, 8, 12; months 6, 9, 12 after infusion of MB-CART2019.1
  Assessment of blood samples for occurrence of B cell aplasia

CONTACTS AND LOCATIONS:
Overall Officials: Peter Borchmann, Prof. Dr., Principal Investigator — University Hospital Cologne
Locations (3):
- Germany (3):
  - Klinikum Augsburg, II. Med. Klinik Haematologie / Onkologie, Augsburg, Bavaria
  - University Hospital Cologne - Department for Internal Medicine I, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Hamburg-Eppendorf, Department of Stem Cell Transplantation, Hamburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Balke-Want H, Godel P, Schmid C, Ayuk FA, Friedrichs B, van Heteren P, Holtkamp S, Zadoyan G, Brillant C, Costa J, Hanssens L, Holzer T, Wohle C, Biedermann S, Burger I, Orentas RJ, Overstijns T, Scheid C, Holtick U, Miltenyi S, Hallek MJ, Borchmann P, Kutsch N. Zamtocabtagene Autoleucel in Relapsed/refractory B-NHL: 5-year Follow Up of a CD20/19 tandem CAR T Cell Phase 1 Trial. Blood Adv. 2026 Jan 9:bloodadvances.2025018073. doi: 10.1182/bloodadvances.2025018073. Online ahead of print. PMID 41512222